CLINICAL TRIAL: NCT04303455
Title: Renin as a Biomarker of Haemodynamic Normalisation: Associations With Outcomes After Cardiac Surgery
Brief Title: Renin as a Biomarker of Haemodynamic Normalisation
Status: Completed | Type: Observational
Sponsor: South West Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Anders Aneman, Professor, South West Sydney Local Health District
Other Study IDs: 2019/PID15341
Record Dates: First submitted 2020-03-08; First posted 2020-03-11 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Shock
Keywords: Biomarkers of shock; Biomarkers of adverse outcomes in shocked patients; Biomarkers of adverse outcomes in cardiothoracic patients
MeSH Terms: conditions — Shock | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: The study will evaluate a cohort of participants meeting the following inclusion criteria:
  1. Admission to ICU after elective and emergency cardiac surgery following cardiopulmonary bypass
  2. Age 18 years and above
  3. Arterial, central venous and pulmonary arterial catheters have been inserted as part of routine care
  Data collection, serum renin among routine blood collection on admission, 6 and 24 hours after admission to ICU
  Interventions: Diagnostic Test: blood sampling

INTERVENTIONS:
Diagnostic Test: blood sampling — sampling serum renin

SUMMARY:
Study design Observational, single centre, prospective cohort study Planned sample size 100 participants

Inclusion criteria The study will evaluate a cohort of participants meeting the following inclusion criteria:

1. admission to the Intensive Care Unit (ICU) after elective and emergency cardiac surgery using cardiopulmonary bypass
2. age 18 years and above
3. arterial, central venous and pulmonary arterial catheters have been inserted as part of routine care Study procedures In addition to routine clinical postoperative data and blood collection, serum renin levels will be analysed on admission, 6 and 24 hours after admission to ICU Study duration 6 months

DETAILED DESCRIPTION:
The renin-angiotensin aldosterone system (RAAS) is integral to cardiovascular homeostasis and involved in the regulation of blood pressure, electrolyte balance and intravascular volume. Renin is produced from the renal juxtaglomerular cells and converts angiotensinogen to angiotensin. Angiotensin is subsequently converted to angiotensin II by angiotensin-converting enzyme (ACE). Angiotensin II also promotes the release of aldosterone.The RAAS has an important role in hypotension to retain water through aldosterone and increase systemic vascular resistance mainly through angiotensin II but also through the release of vasopressin.

The RAAS can become dysregulated in critically ill shocked patients. In states such as septic shock the effects of the RAAS are antagonized through the production of vasodilators such a nitric oxide and both angiotensin I and angiotensin II receptors are down regulated. Activation of angiotensin I receptors may furthermore result in the production of pro-inflammatory cytokines that results in further vasodilation and contributes to cardiovascular compromise.

While the RAAS has been extensively investigated in cardiovascular patients there is a paucity of studies relevant to ICU. A recent study suggested that raised serum renin levels in patients with sepsis is associated with acute renal failure. Another study of a small heterogeneous cohort of critically ill patients compared renin to lactate as marker of tissue perfusion.

As RAAS is closely related to the volume state, there is a physiological rationale to investigate serum renin levels together with variables to monitor the intravascular volume, including assessment of the mean systemic filling pressure (Pmsf). An analogue of the Pmsf will be calculated in this study based on routine postoperative haemodynamic monitoring (mean arterial pressure, MAP, central venous pressure, CVP, cardiac output, CO).

Furthermore, there is no current research which looks at serum renin as marker of hemodynamic normalization or association with outcomes after cardiac surgery which is the main purpose of this study.

Serum renin as a candidate sensitive biomarker of hemodynamic homeostasis will be compared to current clinical markers of resuscitation and perfusion including cardiac index, mixed venous oxygen saturation, lactate and venoarterial carbon dioxide gradients.

If the serum renin concentration is found to be a marker of resuscitation and hemodynamic status, the study will examine any associations with lack of hemodynamic normalization and morbidity in cardiothoracic patients. A pragmatic, composite morbidity outcome at 30 days will be used as the primary endpoint. This includes renal impairment, myocardial infarction, persistent cardiogenic shock, arrythmia, respiratory failure, delirium and stroke. An exploratory, secondary outcome will focus on whether serum renin concentrations are associated with acute kidney injury and the need of renal replacement therapy in post cardiac surgical patients.

ELIGIBILITY:
Inclusion Criteria:

1. Admission to ICU after elective and emergency cardiac surgery following cardiopulmonary bypass
2. Age 18 years and above
3. Arterial, central venous catheters and pulmonary arterial catheters are inserted preoperatively

Exclusion Criteria:

1. Age under 18 years
2. Known pregnancy
3. Arterial, central venous catheters and pulmonary arterial catheters that are not indicated as part of routine care
4. End stage renal disease requiring renal replacement therapy
5. Participants with known Child Pugh A cirrhosis or greater
6. Treatment with any steroids
7. Participant is not expected to live beyond the day after the day of admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Admission to ICU after elective and emergency cardiac surgery following cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2020-03-24 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Patterns of changes in serum renin concentrations are associated with composite morbidity at 30 days in participants who have undergone cardiac surgery. | 30 days

SECONDARY OUTCOMES:
Patterns of changes in serum renin concentrations correlate with current markers of resuscitation in participants who have undergone cardiac surgery ( C.I, SvO2, MAP, urine output, serum lactate, based deficit, venoarterial CO2 gradients) | 24 hours
Serum renin concentrations correlate with Pmsa in postoperative cardiac surgical patients | 24 hours
Patterns of changes in serum renin concentrations are associated with AKI or the need for CRRT in participants who have undergone cardiac surgery | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Wajid Khan, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No
Results of the study will be shared

REFERENCES:
- [Background] Nguyen M, Denimal D, Dargent A, Guinot PG, Duvillard L, Quenot JP, Bouhemad B. Plasma Renin Concentration is Associated With Hemodynamic Deficiency and Adverse Renal Outcome in Septic Shock. Shock. 2019 Oct;52(4):e22-e30. doi: 10.1097/SHK.0000000000001285. PMID 30407370
- [Background] Myles PS. Meaningful outcome measures in cardiac surgery. J Extra Corpor Technol. 2014 Mar;46(1):23-7. PMID 24779115
- [Result] Hall A, Busse LW, Ostermann M. Angiotensin in Critical Care. Crit Care. 2018 Mar 20;22(1):69. doi: 10.1186/s13054-018-1995-z. PMID 29558991
- [Result] Khanna AK. Tissue Perfusion and Prognosis in the Critically Ill-Is Renin the New Lactate? Crit Care Med. 2019 Feb;47(2):288-290. doi: 10.1097/CCM.0000000000003582. No abstract available. PMID 30653057